CLINICAL TRIAL: NCT04819503
Title: Dependency of the Peripheral Nervous System as a Driver for Post-amputation Pain and Therapeutic Effects of Deep Repetitive Transcranial Magnetic Stimulation in a Randomized Double-blind Sham-controlled Study
Brief Title: Mechanisms and Treatment of Post-amputation Neuropathic Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment and technical difficulties
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Nadine Farnes, PhD, Oslo University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 77110
Record Dates: First submitted 2021-03-16; First posted 2021-03-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Neuropathic Pain; Phantom Limb Pain; Amputation
Keywords: repetitive transcranial magnetic stimulation; spinal anaesthesia
MeSH Terms: conditions — Neuralgia; Phantom Limb | interventions — Anesthesia, Spinal; Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: All included patients participate in sub-study 1 and 2. Sub-study 1 is an observational study where patients undergo a spinal anaesthesia in an open label manner. In sub-study 2, patients are once randomly assigned in a 1:1 ratio to one of two counterbalanced arms: either they first receive active rTMS, and then after a 9 week washout period, sham rTMS, or they first receive sham rTMS, and then after 9 weeks of washout, active rTMS. Thus, patients undergo stimulation with deep rTMS in a double blinded randomised controlled trial with a 2 x 2 cross-over design, receiving both active and placebo stimulation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding is achieved by inserting a card into the rTMS stimulator which determines whether the patients receive active or sham stimulation. Thus, both experimenter and patients are blinded towards group allocation. Care providers are also blinded to the treatment allocation.
  The main efficacy analyses will be performed blinded without identification of participants and group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active and then sham repetitive transcranial magnetic stimulation (Other): Deep rTMS is delivered with the Brainsway H7-coil (Brainsway, Jerusalem, Israel) applied via a helmet placed on the head targeting the primary motor cortex of the leg.
  Sham stimulation is delivered with a sham coil placed in the helmet encasing the active rTMS coil. Sham rTMS sessions will use exactly the same parameters of stimulation as active rTMS.
  Interventions: Drug: Spinal anaesthesia (sub-study 1); Device: Repetitive transcranial magnetic stimulation (sub-study 2)
- Sham and then active repetitive transcranial magnetic stimulation (Other): Deep rTMS is delivered with the Brainsway H7-coil (Brainsway, Jerusalem, Israel) applied via a helmet placed on the head targeting the primary motor cortex of the leg.Sham stimulation is delivered with a sham coil placed in the helmet encasing the active rTMS coil. Sham rTMS sessions will use exactly the same parameters of stimulation as active rTMS.
  Interventions: Drug: Spinal anaesthesia (sub-study 1); Device: Repetitive transcranial magnetic stimulation (sub-study 2)

INTERVENTIONS:
Drug: Spinal anaesthesia (sub-study 1) — We will conduct two sub-studies on the same patient group. Sub-study 1 is an observational study where patients with phantom and/or residual limb pain after lower limb amputation will be given spinal anaesthesia with 1% Chloroprocaine in an open label manner to investigate whether the peripheral nervous system is a necessary driver of their pain.
Device: Repetitive transcranial magnetic stimulation (sub-study 2) — After sub-study 1, the same patients will enter sub-study 2 where they are randomly assigned to receive either first active rTMS (10 days over 2 weeks), and then after a 9 week washout period, sham rTMS (10 days over 2 weeks), or they first receive sham rTMS, and then after 9 weeks of washout, active rTMS. Thus, patients undergo stimulation with deep rTMS in a double blinded randomised controlled trial with a 2 x 2 cross-over design, receiving both active and placebo stimulation

SUMMARY:
Phantom and residual limb pain are types of peripheral neuropathic pain that are difficult to treat and where the underlying mechanisms are still not fully understood. Repetitive transcranial magnetic stimulation (rTMS) of the motor cortex is an increasingly studied technique for the treatment of neuropathic pain and has shown modest effects in pain intensity reduction for the treatment of neuropathic pain. Newer rTMS coils provide the opportunity to stimulate larger brain areas, which could provide a better treatment option compared to conventional coils. The aims of this study are to investigate whether the peripheral nervous system is a necessary driver of phantom limb pain and/or residual limb pain in patients with lower limb amputation using spinal anaesthesia, and to assess the analgesic efficacy of deep H-coil rTMS compared to sham stimulation in the same patients.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* Unilateral or bilateral lower limb amputation resulting in residual limb pain and/or phantom pain, fulfilling the criteria for definite neuropathic pain
* Usual pain intensity at least 4/10 over the past 24 hrs using the numerical scale of the BPI at screening
* Daily pain
* Pain for at least 3 months
* Stable pharmacological treatment for pain or no pharmaceutical treatment at least 1 month prior to the study
* Patients who can be followed for the whole duration of the study
* Minimum 4/10 pain intensity at the time of spinal anaesthesia for sub-study 1

Exclusion Criteria:

* Any clinically significant or unstable medical or psychiatric disorder
* Subjects protected by law (guardianship or tutelage measure)
* History of or current substance abuse (alcohol, drugs)
* Pending litigation
* Contraindications to spinal anaesthetic block (e.g. use of prescribed or non-prescribed medication that can increase risk of bleeding such as anticoagulants, non-steroidal anti-inflammatory drugs and acetylsalicylic acid)
* Contraindication to rTMS (past severe head trauma, history of epilepsy or ongoing epilepsy, active cerebral tumour, past neurosurgical intervention, intracranial hypertension, implanted devices not compatible such as cardiac pacemaker and neurostimulator, cochlear implants, pregnancy or lactation. All women of childbearing age will be required to have negative pregnancy test at inclusion and to be using contraception)
* Other pain conditions more severe than phantom and residual limb pain.
* Inability to understand the protocol or to fill out the forms
* Other ongoing research protocol or recent past protocol within one month before the inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Percentage spontaneous pain intensity reduction (sub-study 1) | Maximum reduction during a time interval from 5-60 minutes after spinal anaesthesia
  Measured on an 11-point numerical rating scale (0 %= no pain reduction; 100 % = complete pain reduction).
Change in usual pain intensity over the past 24 hours from baseline to 1 week after each treatment (sub-study 2 | Average of usual pain scores one week before each treatment (baseline week) and 1 week after each treatment
  Usual pain intensity over the past 24 hours is measured on a 11-point numerical rating scale (0 = no pain, 10 = worst pain intensity imaginable of the current pain condition) every day in a diary at the same hour (end of the day). Analgesic efficacy of active and sham treatment is considered the decrease in usual pain intensity scores between the average of each baseline week (one week before treatment) and average of 1 week after last stimulation of each treatment.

SECONDARY OUTCOMES:
Intensity of brush induced allodynia (sub-study 1) | Measured before, 5 minutes and 30 minutes after spinal anaesthesia
  Maximal pain intensity after 3 brush strokes (SOMEDIC brush) to the area of maximal pain with 2 seconds intervals and 3 cm brush strokes lasting 1 second on a 0-10 numerical rating scale (0 = no pain, 10 = worst pain imaginable)
Intensity of pressure induced allodynia (sub-study 1) | Measured before, 5 minutes and 30 minutes after spinal anaesthesia
  Maximal pain intensity after 3 presses using an algometer (10 kPa) to the area of maximal pain with 2 seconds intervals lasting 10 seconds on a 0-10 numerical rating scale (0 = no pain, 10 = worst pain imaginable)
Pin-prick sensitivity (sub-study 1) | Measured before, 5 minutes and 30 minutes after spinal anaesthesia
  Compared to contralateral area, sensitivity is measured with a weighted needle (512 mN) on a 0-10 numerical rating scale where 5 is normal sensation, 0 is no sensation and 10 is maximal painful/intense sensation
Spontaneous pain intensity right now (sub-study 1) | Measured before, and 5, 10, 15, 20, 25, 30, 60, 90 and 120 minutes after spinal anaesthesia
  Measured on a 0-10 numerical rating scale where 0 indicates no pain and 10 indicates worst pain imaginable
Usual pain intensity over the past 24 hours (sub-study 2) | Analgesic efficacy of active and sham treatment is measured as the decrease in pain intensity scores between baseline values (one week before treatment) and 3 weeks after the last stimulation.
  Measured every day in a diary at the same hour (end of the day) on an 11-point numerical rating scale (0 = no pain, 10 = worst pain intensity imaginable of the current pain condition)
Pain intensity (sub-study 2) | Before, 1 week and 3 weeks after the end of each stimulation period
  Pain intensity right now, maximum and minimum pain intensity over the last 24 hours, rated on a numerical rating scale from 0 (no pain) to 10 (pain as bad as you can imagine)
Pain unpleasantness (sub-study 2) | Before, 1 week and 3 weeks after the end of each stimulation period
  Pain unpleasantness right now, maximum, minimum, and usual pain unpleasantness during the last 24 hours, rated in a numerical rating scale from 0 (no pain/unpleasantness) to 10 (unpleasantness as bad as you can imagine)
Pain diary of pain duration, paroxysms and pain interference on sleep (sub-study 2) | Every day 1 week before each stimulation period and up to three weeks after
  Pain duration (percentage wakefulness in pain on an 11-point numerical rating scale; 0% = pain and 100 % = pain all the time), number, duration and usual intensity of pain paroxysms (11-point numerical rating scale; 0 = no pain and 10 = pain as bad as you can imagine), and pain interference on sleep (11-point numerical rating scale; 0 = no interference on sleep, 10 = pain interference on sleep as bad as you can imagine)
Proportion of responders (sub-study 2) | Before,1 week and 3 weeks after the end of each stimulation period
  Proportion of responders with at least 30% and 50% usual pain intensity reduction compared to prestimulation values allowing to calculate Numbers Needed to Treat for 30 % and 50 % pain relief.
Percentage pain intensity reduction (sub-study 2) | Before,1 week and 3 weeks after the end of each stimulation period
  Percentage pain intensity reduction on an 11-point numerical rating scale (0 %= no pain reduction; 100% complete pain reduction)
Pain interference (sub-study 2) | Before,1 week and 3 weeks after the end of each stimulation period
  7 items for pain interference on physical and psychological function from the Brief Pain Inventory rated from 0 (does not interfere), to 10 (complete interference)
Neuropathic Pain Symptom Inventory (sub-study 2) | Before,1 week and 3 weeks after the end of each stimulation period
  Measures mean intensity of 10 neuropathic symptoms during the last 24 hours on 11-point (0-10) numerical scales.
Short form McGill Pain questionnaire (sub-study 2) | Before,1 week and 3 weeks after the end of each stimulation period
  The sensory and affective score of the short form McGill Pain questionnaire which consists of 15 items measured on a 4 point scale.
Hospital Anxiety and Depression Scale (sub-study 2) | Before,1 week and 3 weeks after the end of each stimulation period
  The Hospital Anxiety and Depression Scale includes 14 items scored as anxiety and depression scores, 7 items assessing depression and 7 anxiety
Pain Catastrophizing Scale (sub-study 2) | Before,1 week and 3 weeks after the end of each stimulation period
  Consists of 13 items describing the occurrence of thoughts and feelings that individuals may experience when in pain rated from 0 (not at all) to 4 (all the time).
Patient Global Impression of Change (sub-study 2) | Before,1 week and 3 weeks after the end of each stimulation period
  Consists of 7 items to evaluate the subjective improvement or deterioration (from very much improved to very much deteriorated)
Insomnia Severity Index (sub-study 2) | Before,1 week and 3 weeks after the end of each stimulation period
  Consists of self-rated questions which maps sleep difficulties specific to insomnia on a 5 point Likert scale
Patient-Specific Functional Scale (sub-study 2) | Before,1 week and 3 weeks after the end of each stimulation period
  The Patient-Specific Functional Scale is a numeric rating scale that measures individually chosen functions that are inhibited by the pain. Patients rate from 0 (unable to perform activity) to 10 (able to perform activity)
Executive functioning using the CANTAB battery | Before,1 week and 3 weeks after the end of each stimulation period
  Composite score and individual scores of the paired associates learning test, stop signal task, spatial working memory test and the multitasking test
Side-effects (sub-study 2) | Immediately after the first rTMS session for both stimulation periods, before and after all other rTMS sessions, and 1 week and 3 weeks after each stimulation period
  Side effects using a specific side effects questionnaire specifically designed for assessment of safety in rTMS studies
Blinding (sub-study 2) | 3 weeks after the end of each stimulation period
  blinding questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Audun Stubhaug, DMedSci, Study Director — Oslo University Hospital
Locations (1):
- Department of Pain Management and Research, Oslo University Hospital and Faculty of Medicine, University of Oslo,, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data collected during the trial will be available to other researchers who provide a methodologically sound proposal, and who adhere to institutional guidelines.
Supporting Information: Study Protocol, ICF
Time Frame: All the individual participant data collected during the trial will be available after deidentification, beginning 3 months and lasting 5 years after publication.
Access Criteria: Requestors will need to sign a data access agreement.